CLINICAL TRIAL: NCT03596476
Title: Diagnostic Yield of Post PRandial Esophageal High Resolution Impedance Manometry in Patients With Gastro-Esophageal Reflux Disease Symptoms Resistant to Proton Pump Inhibitor Therapy
Acronym: PRIMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0043; 2018-A01591-54 (Other: ID-RCB)
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Gastro-esophageal Reflux Disease
Keywords: Gastro-esophageal reflux; High resolution Impedance Manometry; Resistance to proton pump inhibitors (PPI)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with persistent GERD (Experimental): Patients with persistent GERD suggestive symptoms despite PPI therapy. All the patients will undergo an upper gastrointestinal (GI) endoscopy, a wireless pH monitoring and a post prandial esophageal High Resolution Impedance Manometry (HRIM). Optional: 24-h pH-impedance monitoring on PPI
  Interventions: Procedure: Upper gastrointestinal (GI) endoscopy; Procedure: Wireless pH monitoring; Procedure: Post prandial esophageal High Resolution Impedance Manometry; Procedure: pH-impedance monitoring

INTERVENTIONS:
Procedure: Upper gastrointestinal (GI) endoscopy — An upper gastrointestinal (GI) endoscopy will be performed at V1. Four esophageal biopsies will be taken in both the proximal and the distal esophagus.
Procedure: Wireless pH monitoring — Wireless pH monitoring will be performed at V1. The pH capsule will be clipped into the esophagus during the upper GI endoscopy. The esophageal pH will be recorded for 96 hours (ambulatory recording).
Procedure: Post prandial esophageal High Resolution Impedance Manometry — Post prandial esophageal HRIM will be performed at V2. The recording will be started after transnasal insertion of the HRIM probe. A standardized meal will be given to the patient (Big Mac, medium portion of French fries, orange juice). The recording will be realized for one hour after the end of the meal.
Procedure: pH-impedance monitoring — 24-h pH-impedance monitoring on PPI will be performed at V3. A transnasal catheter will be inserted into the esophagus and the recording will be performed for 24 hours (ambulatory recording).

SUMMARY:
Gastro-esophageal reflux disease (GERD) is defined as the reflux of gastric content into the esophagus that causes troublesome symptoms or complications. Nine to 30% of the population suffers from GERD-suggestive symptoms (heartburn, regurgitation, chest pain, chronic couch, sore throat). In the absence of warning signs, proton pump inhibitors (PPI) are prescribed as first-line treatment. However, 20 to 60% of patients are unsatisfied because of persistent symptoms when taking PPI. Causes of persistent symptoms are: erroneous diagnosis of GERD (up to 50% of PPI non-responders), rumination syndrome, excessive weakly acid reflux on PPI due to defective esophago-gastric junction or an excessive number of transient lower esophageal sphincter relaxations (main mechanism of GERD), poor acid secretion inhibition on PPI, and non-compliance to therapy. Complementary examinations are indicated to explain persistent GERD symptoms. Upper gastro-intestinal endoscopy is performed first to rule out an esophageal tumor and to identify erosive esophagitis, a specific sign of GERD. However, it is normal in up to 70% of symptomatic GERD patients. Direct detection of reflux episodes is then requested to confirm GERD. The gold standard for reflux detection is the ambulatory measurement of esophageal pH for 24 to 96 hours using a catheter (catheter-based pH-monitoring) or a capsule clipped into the esophagus (wireless pH-monitoring). Reflux episodes are defined as an esophageal pH < 4. Another method of reflux detection is based on liquid and gas detection in the esophagus using pH-impedance monitoring. Recently the combination of impedance and esophageal pressure monitoring, called esophageal high resolution impedance manometry (HRIM) was introduced to simultaneously identify reflux episodes and their mechanisms. It has several advantages over esophageal pH measurement: shorter recording duration (1 or 2 hours post prandial) and identification of reflux mechanisms that might guide the choice of the best therapeutic option.

Hypothesis: The 1-hour post prandial esophageal HRIM might be useful to diagnose GERD.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Typical symptoms of GERD (heartburn, regurgitation) at least twice a week despite PPI therapy for at least one month.
* Reflux Disease Questionnaire (RDQ) score off PPI > 3
* Subject with health insurance

Exclusion Criteria:

* Previous esophago-gastric surgery,
* Previous history of developing esophageal or gastric tumor, esophageal stricture, or esophageal varices
* Pregnancy (assessment at V0)
* Contraindication to general anesthesia,
* Contraindications to the wireless capsule pH-monitoring: pacemakers, implantable cardiac defibrillator,
* Contraindications to HRIM: inability to tolerate nasal intubation, significant bleeding disorders for which nasal intubation is contraindicated, known esophageal obstruction is preventing the passage of the HRIM probe.
* Intolerance or allergy to one component of the test meal,
* Intolerance or allergy to PPI,
* Inability to give consent,
* Mentally unbalanced patients, under supervision or guardianship
* Decline to participate in the study,
* Participation in another study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Number of reflux episodes identified on the post prandial HRIM | 1 hour after the end of the meal
  The diagnostic performance of the number of reflux episodes measured by 1-hour post prandial HRIM will be evaluated by estimating the Area Under the ROC Curve and its 95% confidence interval. The gold standard to define GERD will be based on esophageal pH measurements with capsule (GERD is defined as acid exposure time (AET; percentage of total time with esophageal pH < 4) greater than 6% for at least one day on wireless pH monitoring).

SECONDARY OUTCOMES:
Acid exposure time measured on wireless pH-monitoring | 4 days
  The diagnosis of GERD based on pH-monitoring. The diagnosis of GERD is positive if acid exposure time (AET; percentage of total time with esophageal pH < 4) is greater than 6% for at least one day on wireless pH monitoring. The diagnosis of GERD is negative (ie absence of GERD) if the AET is below 4% during the 4 days of wireless monitoring. In the other instance , the diagnosis of GERD is uncertain.
Reflux mechanisms defined on post prandial HRIM | 1 hour after the end of the meal
  Description of the reflux mechanisms associated with reflux episodes: rumination, transient lower esophageal sphincter relaxation (TLESR), defective esophago-gastric junction (EGJ) or unknown.
Baseline impedance measured on post prandial HRIM | 1 hour after the end of the meal
  Measure of baseline impedance on a period without swallow 3 and 5 cm above the proximal border of the esophago-gastric junction
Resting pressure of the esophago-gastric junction | 1 hour
  Measure of the resting pressure of the esophago-gastric junction on a period without swallowing
Esophageal histology | 4 weeks
  Presence of eosinophils cells in the esophageal mucosa > 15/hpf, dilated intercellular spaces, and/or papillar elongation
Response to 4-week regimen of dose PPI | 4 weeks
  Clinical response is defined as a Reflux Disease Questionnaire score on PPI ≤ 3 after 4-week treatment
Normalization of the number of reflux episodes detected on 24-h pH-impedance monitoring performed on PPI | 1 day
  The number of reflux episodes is normalized if the total number of reflux episodes is < 60 /24 h) on pH-impedance monitoring performed on PPI.
Normalization of the acid exposure time measured on 24-h pH-impedance monitoring performed on PPI | 1 day
  The esophageal acid exposure (AET) is normalized if it is below 4% on pH-impedance monitoring performed on PPI.
Patient's preference regarding the type of examination | 1 day
  Percentage of patients who preferred the wireless pH capsule and percentage of patients who preferred HRIM.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service d'Hepato-Gastroenterologie - Hôpital Trousseau - CHU de Tours, Chambray-lès-Tours
  - Service d'Hepato-Gastroenterologie - Hôpital Louis Mourier - APHP, Colombes
  - Service d'Explorations Fonctionnelles Digestives - Hôpital Edouard Herriot - HCL, Lyon
  - Service d'Hepato-Gastroenterologie - Hôtel Dieu - CHU de Nantes, Nantes
  - Service d'Hepato-Gastroenterologie - Hôpital Haut Lévêque - CHU de Bordeaux, Pessac
  - Service d'Hepato-Gastroenterologie - Hôpital Pontchaillou- CHU de Rennes, Rennes
  - Service de Physiologie Digestive, Respiratoire, Urinaire et Sportive - CHU de Rouen, Rouen